CLINICAL TRIAL: NCT04899700
Title: Linked Color Imaging vs. High-definition White Light Endoscopy for the Evaluation of Post-polypectomy Scars of Non-pedunculated Polyps. A Randomized Controlled Cross-over Trial. (LCI-Scar Study).
Brief Title: Linked Color Imaging Versus White Light Endoscopy for the Evaluation of Scars of Non-pedunculated Polyps. LCI Scar Study.
Acronym: LCIScar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: European Society of Gastrointestinal Endoscopy (Other)
Responsible Party: Principal Investigator, María Pellisé, María Pellisé, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: HCB/2020/0076
Record Dates: First submitted 2020-11-12; First posted 2021-05-24 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Polyp of Colon
Keywords: postpolypectomy scar; Linked color imaging
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Intervention Model Description: Colonoscopy will be performed in tandem by two different endoscopist.
  Patients will be randomized to two groups:
  * WLE-LCI
  * LCI-WLE
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WLE-LCI (Placebo Comparator): First endoscopist will perform an optical diagnosis of recurrence of post-polypectomy scar with WLE. Then a second diagnosis will be performed by the same endoscopist with blue light imaging (BLI)
  Interventions: Device: Linked Color Imaging; Other: White light endoscopy
- LCI-WLE (Active Comparator): First endoscopist will perform an optical diagnosis of recurrence of post-polypectomy scar with Linked Color Imaging (LCI). Then a second diagnosis will be performed by the same endoscopist with blue light imaging (BLI)
  Interventions: Device: Linked Color Imaging; Other: White light endoscopy

INTERVENTIONS:
Device: Linked Color Imaging — Inspection of the postpolypectomy scar will be made with Linked Color Imaging
Other: White light endoscopy — Inspection of the postpolypectomy scar will be made with White light Endoscopy

SUMMARY:
Careful inspection and evaluation of the post-polipectomy scars of polyps greater than 20 mm looking for residual polyp is mandatory. LCI has demonstrated to improve polyp and adenoma detection rate in previous studies. However, to our knowledge no previous studies have been made for validation of LCI for optical diagnosis of a scar looking for residual neoplasia after a previous polypectomy. We hypothesize that LCI will improve the optical diagnosis of polyp recurrence compared to WLE. So, our aim is to compare the efficacy of linked color imaging for optical diagnosis of post-polypectomy scar recurrence compared with high-definition white light endoscopy.

DETAILED DESCRIPTION:
Polypectomy is highly effective in reducing cancer risk by resection of colon cancer precursors: adenomas and serrated lesions1. Despite expertise and good technique, up to 20% of non-pedunculated colorectal polyps larger than 20 mm resected by piecemeal endoscopic mucosal resection (EMR) show scar recurrence2. High recurrence rate implies a higher burden of subsequent surveillance and therapeutic colonoscopies, resulting in patient medicalization and increased costs.

Careful inspection and evaluation of the post-polipectomy scars looking for residual polyp is mandatory. In the past few years several techniques have been developed to improve optical diagnosis. One of them, virtual chromoendoscopy have been developed to overcome laboriousness of conventional chromoendoscopy. A recently a well-designed randomized controlled trial has demonstrated the accuracy of high definition white light endoscopy (WLE) and narrow band imaging (NBI) with or without magnification for diagnosis of scar recurrence after an endoscopic mucosal resection3. High diagnostic values were found for all the modalities but the diagnosis accuracy was higher in NBI with near focus. In cases of high confidence, if the optical diagnosis with NBI plus near focus for scar recurrence is negative, no biopsies are needed3. In view of these findings, the European Society of Gastrointestinal Endoscopy (ESGE) recommends the use of virtual or dye-based chromoendoscopy in addition to WLE for the detection of residual neoplasia in the polypectomy scar after a piecemeal resection.

Fujifilm® (HDTV, ELUXEOTM 700 System, Fujifilm® Tokyo, Japan) has developed a new generation of electronic endoscopy system that employs 4 different-wavelength LEDs as light sources. By changing the intensity of each of 4 LEDs, a white light mode and a Linked Color Imaging (LCI) and Blue Light Imaging (BLI) mode can be obtained. The white light mode is similar to conventional endoscopy using a Xenon lamp while LCI and BLI are the new technologies incorporated the system allowing a bright image-enhanced chromoendoscopy. In both BLI and LCI mode, the peak intensity of the LEDs is set at 410nm±10nm. As this is the peak absorption of light of hemoglobin, microvascular structures at the surface of the mucosa can be distinguished more clearly from blood vessels in the deep mucosa. In contrast to BLI, LCI also acquires the white light in an appropriate balance. The acquired color information is reallocated to differentiate the colors close to the mucosal color, i.e. information for several colors is simultaneously expanded so that the reddish and whitish colors become redder and whiter, respectively. Thereby, mucosal surface patterns are better visualized and this could potentially increase the detection of polyps by improving the visibility of colorectal lesions.

LCI has demonstrated to improve polyp and adenoma detection rate in previous studies5-7. However, to our knowledge no previous studies have been made for validation of LCI for optical diagnosis of a scar looking for residual neoplasia after a previous polypectomy. We hypothesize that LCI will improve the optical diagnosis of polyp recurrence compared to WLE. Therefore, the aim of this study is to evaluate the efficacy of LCI for optical diagnosis of post-polypectomy scar recurrence compared with WLE.

ELIGIBILITY:
Inclusion Criteria:

* Any patient ≥18 years undergoing surveillance colonoscopy after a previous polypectomy of one or more non-pedunculated polyps greater than 15 mm.
* Provide informed consent.

Exclusion Criteria:

* Inflamatory bowel disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Number of recurrence on postpolypectomy scars with White light endoscopy | 2 years
Number of recurrence on postpolypectomy scars with LCI | 2 years
Number of recurrence on postpolypectomy scars detected with AI | 2 years

SECONDARY OUTCOMES:
Elapsed time | 2 years

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - María Pellisé. MD. PhD., Barcelona
  - Oswaldo ortiz, Barcelona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kandel P, Brand EC, Pelt J, Ball CT, Chen WC, Bouras EP, Gomez V, Raimondo M, Woodward TA, Wallace MB; EMR SCAR Group. Endoscopic scar assessment after colorectal endoscopic mucosal resection scars: when is biopsy necessary (EMR Scar Assessment Project for Endoscope (ESCAPE) trial). Gut. 2019 Sep;68(9):1633-1641. doi: 10.1136/gutjnl-2018-316574. Epub 2019 Jan 11. PMID 30635409
- [Result] Bisschops R, East JE, Hassan C, Hazewinkel Y, Kaminski MF, Neumann H, Pellise M, Antonelli G, Bustamante Balen M, Coron E, Cortas G, Iacucci M, Yuichi M, Longcroft-Wheaton G, Mouzyka S, Pilonis N, Puig I, van Hooft JE, Dekker E. Advanced imaging for detection and differentiation of colorectal neoplasia: European Society of Gastrointestinal Endoscopy (ESGE) Guideline - Update 2019. Endoscopy. 2019 Dec;51(12):1155-1179. doi: 10.1055/a-1031-7657. Epub 2019 Nov 11. PMID 31711241
- [Result] Moss A, Bourke MJ, Williams SJ, Hourigan LF, Brown G, Tam W, Singh R, Zanati S, Chen RY, Byth K. Endoscopic mucosal resection outcomes and prediction of submucosal cancer from advanced colonic mucosal neoplasia. Gastroenterology. 2011 Jun;140(7):1909-18. doi: 10.1053/j.gastro.2011.02.062. Epub 2011 Mar 8. PMID 21392504
- [Result] Paggi S, Mogavero G, Amato A, Rondonotti E, Andrealli A, Imperiali G, Lenoci N, Mandelli G, Terreni N, Conforti FS, Conte D, Spinzi G, Radaelli F. Linked color imaging reduces the miss rate of neoplastic lesions in the right colon: a randomized tandem colonoscopy study. Endoscopy. 2018 Apr;50(4):396-402. doi: 10.1055/a-0580-7405. Epub 2018 Mar 14. PMID 29539651